CLINICAL TRIAL: NCT07399574
Title: Accuracy, Safety, and Clinical Performance of a Diquat Quantitative Detection Kit (In-Situ Ionization Mass Spectrometry) and a Portable Mass Spectrometry System for Quantifying Diquat Concentrations in Human Blood Samples (Whole Blood/Plasma)
Brief Title: Diagnostic Accuracy of A Diquat Quantitative Detection Kit and A Portable Mass Spectrometry System for Quantifying Diquat Concentrations in Human Blood Samples
Status: Not yet recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hao Sun, Principal Investigator, Clinical Associate Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: 2025-1207-02
Record Dates: First submitted 2026-01-26; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Diquat Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood specimens will be collected from participants, including whole blood and plasma. At least 2 mL of venous blood will be drawn into anticoagulant tubes (heparin sodium or EDTA). Plasma will be separated by centrifugation (approximately 3000×g for 10-15 minutes) when needed. Samples may include qualified residual specimens remaining after routine clinical testing. Fresh specimens will be tested immediately when feasible, or stored at 2-6°C and analyzed within 24 hours, while a subset of samples may be stored at -80°C for frozen-sample comparisons under routine clinical storage conditions.

GROUPS / COHORTS (4):
- Diquat Poisoning Group (Low Concentration): Participants presenting to the emergency department with clinically diagnosed acute diquat poisoning whose diquat concentration is classified into the low concentration stratum.
  Interventions: Device: Portable Mass Spectrometry Analysis System for Quantitative Diquat Detection (with Diquat Quantitative Detection Kit; In-Situ/Ambient Ionization Mass Spectrometry Method)
- Diquat Poisoning Group (Medium Concentration): Participants presenting to the emergency department with clinically diagnosed acute diquat poisoning whose diquat concentration is classified into the medium concentration stratum.
  Interventions: Device: Portable Mass Spectrometry Analysis System for Quantitative Diquat Detection (with Diquat Quantitative Detection Kit; In-Situ/Ambient Ionization Mass Spectrometry Method)
- Diquat Poisoning Group (High Concentration): Participants presenting to the emergency department with clinically diagnosed acute diquat poisoning whose diquat concentration is classified into the high concentration stratum.
  Interventions: Device: Portable Mass Spectrometry Analysis System for Quantitative Diquat Detection (with Diquat Quantitative Detection Kit; In-Situ/Ambient Ionization Mass Spectrometry Method)
- Non-Diquat Poisoning Group (Negative Control): Participants presenting to the emergency department who are not diagnosed with acute diquat poisoning will be enrolled as negative controls. Their blood samples will be tested in parallel to support evaluation of method performance and to confirm negative results in non-diquat cases.
  Interventions: Device: Portable Mass Spectrometry Analysis System for Quantitative Diquat Detection (with Diquat Quantitative Detection Kit; In-Situ/Ambient Ionization Mass Spectrometry Method)

INTERVENTIONS:
Device: Portable Mass Spectrometry Analysis System for Quantitative Diquat Detection (with Diquat Quantitative Detection Kit; In-Situ/Ambient Ionization Mass Spectrometry Method) — The portable mass spectrometry analysis system is an in vitro diagnostic device used with a diquat quantitative detection kit based on an in-situ/ambient ionization mass spectrometry method to quantify diquat concentrations in human blood samples. Whole blood specimens collected in routine clinical care will be analyzed using this device, and the quantitative results will be compared against those obtained using the reference standard method, liquid chromatography-tandem mass spectrometry (LC-MS/MS), to evaluate analytical accuracy and agreement. Each specimen will be tested repeatedly (three measurements per sample), and the mean value will be used for statistical analysis. The study is observational and non-interventional, and test results generated by the portable mass spectrometry system are used for research evaluation purposes and do not alter routine clinical diagnosis or treatment decisions

SUMMARY:
This is an observational, non-interventional diagnostic accuracy study designed to evaluate a diquat quantitative detection kit (ambient ionization mass spectrometry method) and a portable mass spectrometry analysis system for measuring diquat concentrations in human blood samples (whole blood/plasma), using LC-MS/MS as the clinical gold standard for comparison.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with suspected or clinically diagnosed acute diquat poisoning, providing whole blood and/or plasma samples, including qualified residual specimens retained after prior clinical testing when available.
2. The participant or their legally authorized representative can fully understand the study purpose and procedures, voluntarily agrees to participate, and is willing and able to comply with the study requirements.
3. Sample collection is performed according to routine clinical standards, with no apparent ethical concerns related to sample acquisition.

Exclusion Criteria:

1. Abnormal sample appearance, such as visible flocculent material or other gross abnormalities.
2. The participant is unable to provide a specimen, or the specimen does not meet testing requirements.
3. Any participant considered inappropriate for inclusion by the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from patients presenting to the emergency department during the study period. The study population includes individuals with suspected or clinically diagnosed acute diquat poisoning, stratified into low, medium, and high concentration groups (15 participants per group), as well as a negative control group consisting of non-diquat-poisoning patients (15 participants), for a total enrollment of 60 participants.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Bland-Altman agreement | Baseline
  Assesses agreement and bias between the two methods; requires most data points within preset LOA
Correlation coefficient between portable MS and LC-MS/MS | Baseline
  Measures linear association of quantitative results; target orrelation coefficient ≥ 0.95
Relative deviation at medical decision levels | Baseline
  Evaluates clinically acceptable error; target relative deviatio within ±15%

SECONDARY OUTCOMES:
Recovery rate (spiked mixed samples vs fresh samples) | Baseline
  Target recovery 85%-115%
Precision (Coefficient of Variation, CV) | Baseline
  Within-run CV ≤ 10%; between-run CV ≤ 15%

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China